CLINICAL TRIAL: NCT03003338
Title: A Monocenter Randomized Double-blind Placebo-controlled Study to Investigate Neuropsychiatric Manifestations of HCV-infection During and After Treatment With Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir
Brief Title: MHH-HCV-NPM-Neuropsychiatric Manifestations of HCV-infection During and After Treatment With OBV/PTV/r and DSV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The recruitment was stopped prematurely by the sponsor in accordance with the principal investigator because of the difficulties to recruit patients and to achieve the planned numbers of patients within a reasonable time frame.
Sponsor: Hannover Medical School (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MHH-HCV-NPM; 2015-004556-22 (EudraCT Number)
Record Dates: First submitted 2016-07-15; First posted 2016-12-28 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hepatitis C, Chronic
Keywords: chronic HCV Genotype 1b infection; HCV RNA; OBV/PTV/r in combination with DSV; neuropsychiatric manifestations
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OBV/PTV/r with DSV followed by placebo (Experimental): OBV/PTV/r in combination with DSV for 12 weeks followed by 12 weeks matching placebo.
  Interventions: Drug: OBV/PTV/r and DSV; Drug: Placebo to match OBV/PTV/r and DSV
- Placebo followed by OBV/PTV/r with DSV (Experimental): Matching placebo for 12 weeks followed by 12 weeks OBV/PTV/r in combination with DSV.
  Interventions: Drug: OBV/PTV/r and DSV; Drug: Placebo to match OBV/PTV/r and DSV

INTERVENTIONS:
Drug: OBV/PTV/r and DSV — OBV/PTV/r (12.5 mg/ 75 mg/ 50 mg) in combination with DSV (250 mg): Two tablets of OBV/PTV/r in the morning and one tablet of DSV in the morning and one tablet of DSV in the evening orally with a meal without regard to fat or calorie content.
  Other Names: Viekirax and Exviera
Drug: Placebo to match OBV/PTV/r and DSV — Placebo to match OBV/PTV/r and DSV

SUMMARY:
This is a 1:1 randomized double-blind Placebo-controlled moncenter Phase IV study to investigate whether a successful interferon-free treatment of HCV-infection with ombitasvir/paritaprevir/ritonavir (OBV/PTV/r) in combination with dasabuvir (DSV) improves the patients' attention ability as compared to placebo as measured with the Att Test Sum Score change from baseline to week 12. A total of 30 patients with non-cirrhotic genotype 1b HCV infection will be randomly assigned to receive 12 weeks verum followed by 12 weeks Placebo (arm A) versus 12 weeks Placebo followed by 12 weeks verum (arm B). Patients will be followed up for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age ≥18 years
3. Chronic hepatitis C virus infection
4. Fatigue Impact Scale Score (FIS) >45 and a sum score (Att Test Sum Score) >0.4 in the battery of attention tests applied.
5. Female who is:

   * practicing total abstinence from sexual intercourse (minimum 1 complete menstrual cycle)
   * sexually active with female partners only
   * not of childbearing potential, defined as:

     * postmenopausal for at least 2 years (defined as amenorrheic for longer than 2 years, age appropriate, and confirmed by a follicle-stimulating hormone [FSH] level indicating a postmenopausal state), or
     * surgically sterile (defined as bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or has a vasectomized partner (s);
   * of childbearing potential and sexually active with male partner(s):

     * currently using an effective method of birth control at the time of screening and
     * agree to practice highly effective methods of birth control while receiving study drugs and at least one effective method of birth control during the follow-up period (see section 4.3). (Note: Ethinylestradiol-containing hormonal contraceptives, including oral, injectable, implantable, patch and ring varieties, may not be used during study drug treatment.)
6. Females of childbearing potential must have negative results for pregnancy tests performed:

   * at Screening on a serum specimen obtained within 28 days prior to initial study drug administration, and
   * on a urine sample obtained on Study Day 1 (prior to dosing).
7. Males who are not surgically sterile and who are sexually active with female partner(s) of childbearing potential must agree to practice an effective form of birth control (see section 4.3) throughout the course of the study, starting with Study Day 1 and for 30 days after stopping study drug.
8. Subject must be able to comply with the dosing instructions for study drug administration and be able to complete the study schedule of assessments.
9. Body Mass Index (BMI) is > 17 to < 40 kg/m2. BMI is calculated as weight measured in kg divided by the square of height measured in meters (m).
10. Confirmation of chronic genotype 1b HCV infection documented by the following:

    Positive for anti-HCV antibody or HCV RNA at least 6 months before Screening, and positive for HCV RNA and anti-HCV antibody at the time of Screening
11. Per local standard practice, documented results of:

    * Index (APRI) ≤ 2 at Screening, or
    * FibroScan® result of < 12 kPa at Screening or
    * The absence of cirrhosis based on a liver biopsy within the last 36 months.
12. HCV > RNA 1000 IU/ml at Screening
13. Subject must be of generally good health as determined by the Investigator.
14. Subject has not been treated with any investigational drug or device or any commercially available anti-HCV agents within 42 days of the Screening visit.

Exclusion Criteria:

1. Any previous exposure to HCV protease inhibitors, HCV NS5A inhibitors or HCV polymerase inhibitors
2. History of severe, life threatening or other significant sensitivity to any drug.
3. Pregnant or nursing female or male with pregnant female partner
4. Recent (within 6-months prior to study drug administration) history of drug or alcohol abuse that could preclude adherence to the protocol.
5. Infection with hepatitis B virus (HBV; defined as HBsAg-positive) or human immunodeficiency virus (HIV)
6. Use of any medication that are contraindicated for use with OBV/PTV/r and DSV within 2 weeks prior to study drug administration or 10 half-lives of the medication whichever is longer (see SmPC of OBV/PTV/r and DSV and section 4.4).
7. Clinically-significant illness (other than HCV) or any other major medical disorder that, in the opinion of the investigator, may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
8. Positive result of a urine drug screen at the Screening Visit for opiates, barbiturates, amphetamines, cocaine, benzodiazepines, phencyclidine, and propoxyphene.
9. History of uncontrolled seizures, cancer (except basal cell carcinoma of the skin), or uncontrolled diabetes, as defined by a hemoglobin A1C level > 8.0% or other systemic diseases that affect directly the CNS and brain metabolites.
10. Gastrointestinal disorder or post operative condition that could interfere with the absorption of the study drug (for example, gastric bypass or severe ulcerative colitis).
11. Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, autoimmune hepatitis, alcoholic liver disease, Wilson's disease, α1 antitrypsin deficiency, cholangitis)
12. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
13. Clinical hepatic decompensation (i.e., clinical ascites, encephalopathy or variceal hemorrhage).
14. Solid organ transplantation.
15. Significant pulmonary disease or significant cardiac disease.
16. Significant drug allergy (such as anaphylaxis or hepatotoxicity).
17. Contraindications for MRI study
18. Screening laboratory analyses show any of the following abnormal laboratory results:

    * Alanine aminotransferase (ALT) > 10 × upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) > 10 × ULN
    * Calculated creatinine clearance (using CKD-EPI equal) < 30 mL/min
    * Albumin < lower limit of normal (LLN)
    * INR > 1.5
    * Hemoglobin < LLN
    * Platelets < 90,000 cells per mm3
    * Total bilirubin > 2.0 mg/dL
    * HCV RNA levels that are above the upper level of assay quantification
19. Screening ECG with clinically significant abnormalities
20. Consideration by the Investigator, for any reason, that the subject is an unsuitable candidate to receive the study medication
21. Donation or loss of more than 400 ml blood within 2 months prior to Baseline/Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Change in the Attention Test Battery Sum Score (Att Test Sum Score) at week 12 (12 weeks minus baseline) | 12 weeks
  To investigate whether a successful interferon-free treatment of HCV-infection with ombitasvir/paritaprevir/ritonavir (OBV/PTV/r) in combination with dasabuvir (DSV) improves the patients' attention ability as compared to placebo as measured with the Att Test Sum Score change from baseline to week 12.

SECONDARY OUTCOMES:
Efficacy of treatment with OBV/PTV/r in combination with DSV for 12w in patients with chronic genotype 1b HCV infection as measured by the proportion of subjects with sustained viral response at FU 12 after discontinuation of therapy | Baseline and FU12
  To investigate whether a treatment with OBV/PTV/r in combination with DSV for 12 wk in patients with chronic genotype 1b HCV infection is safe and effective in patients with chronic fatigue and impaired neuropsychiatric function
Efficacy of treatment with OBV/PTV/r in combination with DSV for 12w in patients with chronic genotype 1b HCV infection as measured by the proportion of subjects with sustained viral response at FU 24 after discontinuation of therapy | Baseline and FU 24
  To investigate whether a treatment with OBV/PTV/r in combination with DSV for 12 wk in patients with chronic genotype 1b HCV infection is safe and effective in patients with chronic fatigue and impaired neuropsychiatric function
Efficacy of treatment with OBV/PTV/r in combination with DSV for 12w in patients with chronic genotype 1b HCV infection as measured by the proportion of subjects with sustained viral response at FU48 after discontinuation of therapy | Baseline and FU 48
  To investigate whether a treatment with OBV/PTV/r in combination with DSV for 12 wk in patients with chronic genotype 1b HCV infection is safe and effective in patients with chronic fatigue and impaired neuropsychiatric function
Change in FIS at Treatment week 12 after Treatment discontinuation | Baseline and week 12
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves FIS.
Change in FIS at Treatment at 12 weeks of follow-up after Treatment discontinuation | Baseline and 12 weeks of follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves FIS.
Change in FIS at Treatment at 24 weeks of follow-up after Treatment discontinuation | Baseline and 24 weeks of follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves FIS.
Change in FIS at Treatment at 48 weeks of follow-up after Treatment discontinuation | Baseline and 48 weeks of follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves FIS.
Change in Repeatable Battery for the Assessment of Neuropsychological Function (RBANS) total score at Treatment week 12 after Treatment discontinuation | Baseline and 12 weeks
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves Repeatable Battery for the Assessment of Neuropsychological Function (RBANS) score.
Change in Repeatable Battery for the Assessment of Neuropsychological Function (RBANS) total score at 12 weeks follow-up after Treatment discontinuation | Baseline and 12 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves Repeatable Battery for the Assessment of Neuropsychological Function (RBANS) score.
Change in Repeatable Battery for the Assessment of Neuropsychological Function (RBANS) total score at 24 weeks follow-up after Treatment discontinuation | Baseline and 24 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves Repeatable Battery for the Assessment of Neuropsychological Function (RBANS) score.
Change in Repeatable Battery for the Assessment of Neuropsychological Function (RBANS) total score at 48 weeks follow-up after Treatment discontinuation | Baseline and 48 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves Repeatable Battery for the Assessment of Neuropsychological Function (RBANS) score.
Change in TAP Attention test scores at Treatment week 12 after Treatment discontinuation | Baseline and 12 weeks
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves TAP Attention test scores.
Change in TAP Attention test scores at 12 weeks of follow-up after Treatment discontinuation | Baseline and 12 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves TAP Attention test scores.
Change in TAP Attention test scores at 24 weeks of follow-up after Treatment discontinuation | Baseline and 24 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves TAP Attention test scores.
Change in TAP Attention test scores at 48 weeks of follow-up after Treatment discontinuation | Baseline and 48 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves TAP Attention test scores.
Change in word-figure Memory test scores for verbal and figural Memory function at Treatment week 12 after Treatment discontinuation | Baseline and 12 weeks
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves word-figure Memory test scores for verbal and figural Memory function.
Change in word-figure Memory test scores for verbal and figural Memory function at 12 weeks of follow-up after Treatment discontinuation | Baseline and 12 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves word-figure Memory test scores for verbal and figural Memory function.
Change in word-figure Memory test scores for verbal and figural Memory function at 24 weeks of follow-up after Treatment discontinuation | Baseline and 24 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves word-figure Memory test scores for verbal and figural Memory function.
Change in word-figure Memory test scores for verbal and figural Memory function at 48 weeks of follow-up after Treatment discontinuation | Baseline and 48 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves word-figure Memory test scores for verbal and figural Memory function.
Change in brain metabolite Levels after anti-viral Treatment | Baseline and 12 weeks
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection results in changes of the cerebral metabolites N-acetyl-aspartate, total creatine, choline, Glutamin/Glutamate, and myo-inositol.
Change in brain metabolite Levels after 12 weeks follow-up | Baseline and 12 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection results in changes of the cerebral metabolites N-acetyl-aspartate, total creatine, choline, Glutamin/Glutamate, and myo-inositol.
Change in brain metabolite Levels after 24 weeks follow-up | Baseline and 24 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection results in changes of the cerebral metabolites N-acetyl-aspartate, total creatine, choline, Glutamin/Glutamate, and myo-inositol.
Change in brain metabolite Levels after 48 weeks follow-up | Baseline and 48 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection results in changes of the cerebral metabolites N-acetyl-aspartate, total creatine, choline, Glutamin/Glutamate, and myo-inositol.
Change in the patients mood at Treatment week 12 | Baseline and week 12
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves the patients mood as measured with the Hospital Anxiety and Depression Score.
Change in the patients mood at 12 weeks follow-up | Baseline and 12 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves the patients mood as measured with the Hospital Anxiety and Depression Score.
Change in the patients mood at 24 weeks follow-up | Baseline and 24 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves the patients mood as measured with the Hospital Anxiety and Depression Score.
Change in the patients mood at 48 weeks follow-up | Baseline and 24 weeks follow-up
  To investigate whether treatment with OBV/PTV/r in combination with DSV for 12 weeks in patients with chronic genotype 1b HCV infection improves the patients mood as measured with the Hospital Anxiety and Depression Score.
Change in the Att Test Sum Score at 12 weeks of follow-up | Baseline and 12 weeks follow-up
Change in the Att Test Sum Score at 24 weeks of follow-up | Baseline and 24 weeks follow-up
Change in the Att Test Sum Score at 48 weeks of follow-up | Baseline and 48 weeks follow-up

OTHER OUTCOMES:
HCV-specific T cell responses | Baseline and 48 weeks follow-up
  To assess any relationship between HCV-specific T cell responses and regulatory T cells
HCV-specific T cell responses | Baseline and 48 weeks follow-up
  To assess any relationship between HCV-specific T cell responses and neuropsychatric symptoms
Relationship between NK cell phenotype and function | Baseline and 48 weeks follow-up
  To assess any relationship between NK cell phenotype and function
Relationship between NK cell phenotype and neuropsychatric symptoms | Baseline and 48 weeks follow-up
  To assess any relationship between NK cell phenotype and neuropsychiatric symptoms
Causality between microbiome composition of the gut and the stage of HCV infection/ liver disease in relation to neuropsychiatric findings | Baseline and 48 weeks follow-up
  To assess causalities between the microbiome composition of the gut and the stage of HCV infection/ liver disease in relation to neuropsychiatric findings

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Wedemeyer, Prof. Dr., Principal Investigator — Hannover Medical School, Department of Gastroenterology, Hepatology and Endocrinology, Carl-Neuberg-Str. 1, 30625 Hannover, Germany
Locations (1):
- Hannover Medical School, Hanover, Germany